CLINICAL TRIAL: NCT06029179
Title: Sodium Zirconium Cyclosilicate Versus Sodium Polystyrene Sulfonate for Treatment of Hyperkalemia in Hemodialysis Patients: A Randomized Clinical Trial
Brief Title: SZC Versus SPS for Treatment of Hyperkalemia in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hyperkalemia treatment in HD
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Hyperkalemia
Keywords: Hyperkalemia; Hemodialysis; Sodium Zirconium Cyclosilicate; Sodium Polystyrene Sulfonate
MeSH Terms: conditions — Hyperkalemia | interventions — sodium zirconium cyclosilicate; polystyrene sulfonic acid

STUDY DESIGN:
Intervention Model Description: This research is a prospective randomized multicentric clinical trial in which 120 hemodialysis patients will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
  * Group A: 60 patients will receive sodium zirconium cyclosilicate (SZC) 5 g once daily on non-dialysis days (15 gm/week) for 8 weeks.
  * Group B: 60 patients will receive sodium polystyrene sulfonate 15 g once daily on non-dialysis days (45 gm/week) for 8 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): 60 patients will receive sodium zirconium cyclosilicate (SZC)
  Interventions: Drug: sodium zirconium cyclosilicate (SZC)
- Group B (Active Comparator): 60 patients will receive sodium polystyrene sulfonate
  Interventions: Drug: sodium polystyrene sulfonate

INTERVENTIONS:
Drug: sodium zirconium cyclosilicate (SZC) — 60 patients will receive sodium zirconium cyclosilicate (SZC) 5 g once daily on non-dialysis days (15 gm/week) for 8 weeks.
  Arms: Group A
Drug: sodium polystyrene sulfonate — 60 patients will receive sodium polystyrene sulfonate 15 g once daily on non-dialysis days (45 gm/week) for 8 weeks.
  Arms: Group B

SUMMARY:
This study aims to compare the effects of Sodium Zirconium Cyclosilicate versus Sodium Polystyrene Sulfonate for treatment of hyperkalemia in patients undergoing regular hemodialysis.

DETAILED DESCRIPTION:
Patients maintained on regular hemodialysis (HD) have a high risk of hyperkalemia (>5.0 mmol/l). Hyperkalemia is a critical medical condition that can result in arrhythmias and sudden cardiac death. Treatment of hyperkalemia in HD patients is challenging.

Therapeutic options for the treatment of hyperkalemia in HD population include potassium binding resins, such as sodium polystyrene sulfonate (SPS), patiromer, and sodium zirconium cyclosilicate. There is limited data about the use of these agents in HD.

ELIGIBILITY:
Inclusion Criteria:

1. ≥3 month of maintenance hemodialysis, 3 times per week for 4 hours.
2. Adult patients with age above 18 years.
3. baseline serum potassium level >5 mEq/L.

Exclusion Criteria:

1. Gastrointestinal diseases (constipation, bleeding, Hx of endoscopy, chronic diarrhea or diarrhea in the past month, malabsorption, GIT surgery, ischemic colitis, necrosis, perforation, ….).
2. Breast feeding or pregnancy.
3. Patients who receive medications to treat hyperkalemia 2 weeks before study.
4. myocardial infarction, acute coronary syndrome, stroke, seizure, or thromboembolic event within 8 weeks before study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Change in serum potassium | 8 weeks
  By assessing serum K at baseline, 24 hrs after first dose, then weekly after the long interdialytic interval

SECONDARY OUTCOMES:
Change in interdialytic weight | 8 weeks
  By assessing change in interdialytic weight
Gastrointestinal side effects | 8 weeks
  By reporting any GIT SE
Change in Blood pressure | 8 weeks
  systolic and diastolic Blood pressure change
Serious adverse events | 8 weeks
  By reporting any serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; Marwa Ahmed Abdelrahman, MD, Study Chair — consultant; Mohamed Aly Abdelhalim, MD, Study Chair — Lecturer
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yusuf AA, Hu Y, Singh B, Menoyo JA, Wetmore JB. Serum Potassium Levels and Mortality in Hemodialysis Patients: A Retrospective Cohort Study. Am J Nephrol. 2016;44(3):179-86. doi: 10.1159/000448341. Epub 2016 Sep 3. PMID 27592170
- [Background] Hoppe LK, Muhlack DC, Koenig W, Carr PR, Brenner H, Schottker B. Association of Abnormal Serum Potassium Levels with Arrhythmias and Cardiovascular Mortality: a Systematic Review and Meta-Analysis of Observational Studies. Cardiovasc Drugs Ther. 2018 Apr;32(2):197-212. doi: 10.1007/s10557-018-6783-0. PMID 29679302
- [Background] Beccari MV, Meaney CJ. Clinical utility of patiromer, sodium zirconium cyclosilicate, and sodium polystyrene sulfonate for the treatment of hyperkalemia: an evidence-based review. Core Evid. 2017 Mar 23;12:11-24. doi: 10.2147/CE.S129555. eCollection 2017. PMID 28356904
- [Background] Fried L, Kovesdy CP, Palmer BF. New options for the management of chronic hyperkalemia. Kidney Int Suppl (2011). 2017 Dec;7(3):164-170. doi: 10.1016/j.kisu.2017.09.001. Epub 2017 Nov 17. PMID 30675431
- [Derived] Elsayed MM, Abdelrahman MA, Sorour AM, Rizk IG, Hassab MAA. Sodium zirconium cyclosilicate versus sodium polystyrene sulfonate for treatment of hyperkalemia in hemodialysis patients: a randomized clinical trial. BMC Nephrol. 2025 May 6;26(1):227. doi: 10.1186/s12882-025-04129-9. PMID 40329202